CLINICAL TRIAL: NCT04930731
Title: Risk Factors and Characteristics of COVID 19 Infection in Patients With Haematological Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ayah Ibrahim Nemr, Resident doctor at haematology unit ,, internal medicine department ,, assiut university, Assiut University
Other Study IDs: COVID 19 &haematological pts
Record Dates: First submitted 2020-09-28; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Covid19
Keywords: Haematological diseases
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. assessment of risk factor of covid 19 in haematological patients
2. assessment of characteristics of covid 19 in haematological patients

DETAILED DESCRIPTION:
An ongoing outbreak of pneumonia associated with a novel coronavirus, severe acute respiratory syndrome (SARS) coronavirus 2, was reported in Wuhan, Hubei Province, China, in December 2019 .

In the following weeks, infections spread across China and other countries around the world .

The Chinese public health, clinical, and scientific communities took action to allow for timely recognition of the new virus and shared the viral gene sequence to the world .

On January 30, 2020, the World Health Organization (WHO) declared the outbreak a Public Health Emergency of International Concern

. On February 12, 2020, the WHO named the disease caused by the novel coronavirus "coronavirus disease 2019" (COVID-19) .

A group of international experts, with a range of specializations, have worked with Chinese counterparts to try to contain the outbreak .

Preliminary reports suggest that patients with an underlying malignancy have inferior outcomes.

While haematology patients are thought to be at increased risk of developing severe complications both due to immune dysfunction from their underlying haematological disorder and immunosuppressive therapies used for treatment, delays in treatment of the underling malignancy may compromise patient safety and survival. Data from other cohorts worldwide suggest mortality from COVID-19 is higher in haematology patients compared to the general population, with reported mortality rates between 39% and 50% in other British haematology patient cohorts.

In particular, a recent UK case series reported significantly higher case fatality rates in haematology patients receiving immunosuppressive or cytotoxic therapy within three months of COVID-19 diagnosis, raising concerns about the delivery of systemic anti-cancer therapy (SACT) during the pandemic.

There is an ongoing need to share collective experience regarding the clinical course of COVID-19 in patients with haematological disorders, particularly regarding implications for SACT delivery, in order to enable patients to receive treatment in a timely and safe manner during the pandemic.

ELIGIBILITY:
Inclusion Criteria:

* patients with haematological diseases who suspected or confirmed to COVID 19 infection..
* patients with age more than 18 years old

Exclusion Criteria:

* patients under the age of 18.
* Patients who refuse to contribute in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 2 groups Group A control group Group B study group
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Risk Factors and Characteristics of COVID 19 infection in Patients with Haematological Diseases | From September 2021 to June 2022
  To identify risk factors and characteristics of COVID 19 in patients with haematological diseases

CONTACTS AND LOCATIONS:
Overall Officials: Safaa A Ahmed, Study Chair — safaakhaled2003@gmail.com

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Blimark C, Holmberg E, Mellqvist UH, Landgren O, Bjorkholm M, Hultcrantz M, Kjellander C, Turesson I, Kristinsson SY. Multiple myeloma and infections: a population-based study on 9253 multiple myeloma patients. Haematologica. 2015 Jan;100(1):107-13. doi: 10.3324/haematol.2014.107714. Epub 2014 Oct 24. PMID 25344526
- [Background] Hilal T, Gea-Banacloche JC, Leis JF. Chronic lymphocytic leukemia and infection risk in the era of targeted therapies: Linking mechanisms with infections. Blood Rev. 2018 Sep;32(5):387-399. doi: 10.1016/j.blre.2018.03.004. Epub 2018 Mar 16. PMID 29571669
- [Background] Chemaly RF, Ghosh S, Bodey GP, Rohatgi N, Safdar A, Keating MJ, Champlin RE, Aguilera EA, Tarrand JJ, Raad II. Respiratory viral infections in adults with hematologic malignancies and human stem cell transplantation recipients: a retrospective study at a major cancer center. Medicine (Baltimore). 2006 Sep;85(5):278-287. doi: 10.1097/01.md.0000232560.22098.4e. PMID 16974212
- [Background] Pinana JL, Gomez MD, Montoro J, Lorenzo I, Perez A, Gimenez E, Gonzalez-Barbera EM, Carretero C, Guerreiro M, Salavert M, Sanz G, Hernandez-Boluda JC, Borras R, Sanz J, Solano C, Navarro D. Incidence, risk factors, and outcome of pulmonary invasive fungal disease after respiratory virus infection in allogeneic hematopoietic stem cell transplantation recipients. Transpl Infect Dis. 2019 Oct;21(5):e13158. doi: 10.1111/tid.13158. Epub 2019 Sep 3. PMID 31402532
- [Background] Whimbey E, Englund JA, Couch RB. Community respiratory virus infections in immunocompromised patients with cancer. Am J Med. 1997 Mar 17;102(3A):10-8; discussion 25-6. doi: 10.1016/s0002-9343(97)80004-6. PMID 10868137